CLINICAL TRIAL: NCT00823563
Title: Evaluation of Patients With Angina in the Absence of Obstructive Coronary Artery Disease
Brief Title: Evaluation of Patients With Non-obstructive Coronary Arteries
Acronym: noCAD
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jennifer A Tremmel, MD, MS, Associate Professor, Stanford University
Other Study IDs: 51267
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Chest Pain; Ischemia
MeSH Terms: conditions — Chest Pain; Ischemia | interventions — Ultrasonography, Interventional

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: 30 cc blood draw
Procedure: Intravascular ultrasound (IVUS)
Procedure: Coronary pressure/flow wire testing
Procedure: Coronary pressure/flow testing: Acetycholine challenge
Procedure: Procedure: Coronary pressure/flow testing: Nitroglycerin challenge
Procedure: Procedure: Procedure: Coronary pressure/flow testing: Adenosine challenge

SUMMARY:
Patients with angina and non-obstructive CAD are common within clinical practice, but remain a challenge with regard to diagnosis and treatment. When these patients undergo a comprehensive evaluation at the time of invasive coronary angiography, occult coronary abnormalities are frequently found. We hope to learn the overall prevalence and presentation of these occult coronary abnormalities and its long term outcome in this patient population.

DETAILED DESCRIPTION:
This is a prospective registry of patients with chest pain, chest discomfort, breathlessness who do not have a blockage in their heart artery. This condition is known as angina/ischemia and non-obstructive coronary arteries (ANOCA/INOCA). The purpose of this registry is to help us understand the prevalence, causes of these conditions, identify effective diagnostic strategy, and long term outcome in this patient population.

Patients will undergo comprehensive invasive evaluation including coronary angiography, intravascular imaging, and physiologic measurements as a standard of care. Details regarding the participant's angiogram, endothelial function testing, microvascular testing, intravascular ultrasound, and myocardial bridge testing, if performed, will be entered into a research database.

Participants may be contacted by email or phone periodically for follow-up information, such as surveys, an update on medical history, and/or a check on their medical status or symptoms. We anticipate gathering these data at 6 months, 1 year, 3 years, 5 years, and 10 years, and every 5 years thereafter following their enrollment.

The overall objective of this registry study is to identify specific endotypes of ANOCA by invasive evaluation and study long term outcome.

Specific goals include:

1. Describe the prevalence of the following ANOCA endotypes: endothelial dysfunction, microvascular dysfunction, vasospastic angina, myocardial bridging (MB), and other disorders of coronary physiology, and non-cardiac chest pain;
2. Characterize the natural history and outcomes of patients with ANOCA and determine variables associated with major adverse cardiovascular events

ELIGIBILITY:
Inclusion Criteria:

1. Patient referred for elective coronary angiography because of a reasonable clinical suspicion of coronary ischemia.
2. Presence of angina or an anginal equivalent (including chest, back, shoulder, arm, neck, jaw discomfort, or shortness of breath brought on by physical exertion, emotional stress, or certain times of day/month).

Exclusion Criteria:

1. Asymptomatic (such as a pre-op cath)
2. Status-post heart transplant
3. Age <18
4. Renal insufficiency (creatinine >1.5)
5. Presence of an acute coronary syndrome (STEMI or NSTEMI), Tako-tsubo, an abnormal ejection fraction (EF<55%), cardiogenic shock, or recent VT/VF
6. Presence of another likely explanation of chest pain, such as pulmonary hypertension or aortic stenosis
7. History of adverse reaction to any of the medications being used (acetylcholine, nitroglycerin, adenosine, or heparin)
8. Currently taking vasoactive medication (such as nitroglycerin)
9. Inability to provide an informed consent, including an inability to speak, read, or understand English, Spanish, Chinese, Farsi, Japanese, Korean, Russian, or Vietnamese
10. A hearing impairment that won't allow for a typical verbal conversation or a visual impairment that won't allow for reading of the written consent
11. Participation in another study (with the exception of the Stanford Gene-PAD study)
12. A potentially vulnerable subject (including minors, pregnant women, economically and educationally disadvantaged, decisionally impaired, and homeless people)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult women and men with angina who have been referred for an elective coronary angiogram because of a reasonable clinical suspicion of coronary ischemia.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2007-06 (Actual); Primary Completion 2047-06 (Estimated); Study Completion 2047-06 (Estimated)

PRIMARY OUTCOMES:
Sex Differences in Endothelial Dysfunction, Microvascular Dysfunction, and Diffuse Plaque | Day of procedure (study day one)
  This outcome is to measure the prevalence of angina and non-obstructive coronary arteries (ANOCA) endotypes
Number of participants with major adverse cardiovascular events (MACE) | 15 years
  MACE - death, heart attack, revascularization, stroke

SECONDARY OUTCOMES:
Change in Seattle angina questionnaire score | Baseline, 6 months, 1 year, 3 year, every 5 years thereafter
  Scores range from 0 - 100, higher score means better outcome
Number of patients with cardiovascular rehospitalization | 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Tremmel, MD, MS, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Background] Tremmel JA, Yeung AC. Ischemic heart disease in women: an appropriate time to discriminate. Rev Cardiovasc Med. 2007 Spring;8(2):61-8. PMID 17603424
- [Background] Rogers IS, Tremmel JA, Schnittger I. Myocardial bridges: Overview of diagnosis and management. Congenit Heart Dis. 2017 Sep;12(5):619-623. doi: 10.1111/chd.12499. Epub 2017 Jul 3. PMID 28675696
- [Background] Pargaonkar VS, Kobayashi Y, Kimura T, Schnittger I, Chow EKH, Froelicher VF, Rogers IS, Lee DP, Fearon WF, Yeung AC, Stefanick ML, Tremmel JA. Accuracy of non-invasive stress testing in women and men with angina in the absence of obstructive coronary artery disease. Int J Cardiol. 2019 May 1;282:7-15. doi: 10.1016/j.ijcard.2018.10.073. Epub 2018 Oct 23. PMID 30527992
- [Background] Lee BK, Lim HS, Fearon WF, Yong AS, Yamada R, Tanaka S, Lee DP, Yeung AC, Tremmel JA. Invasive evaluation of patients with angina in the absence of obstructive coronary artery disease. Circulation. 2015 Mar 24;131(12):1054-60. doi: 10.1161/CIRCULATIONAHA.114.012636. Epub 2015 Feb 20. PMID 25712205
- [Background] Tremmel JA, Schnittger I. Myocardial bridging. J Am Coll Cardiol. 2014 Nov 18-25;64(20):2178-9. doi: 10.1016/j.jacc.2014.07.993. Epub 2014 Nov 10. No abstract available. PMID 25457408
- [Background] Tremmel JA. To Define Is to Limit: Is That Good or Bad When it Comes to Chest Pain? JACC Cardiovasc Interv. 2016 Mar 28;9(6):562-4. doi: 10.1016/j.jcin.2016.02.002. Epub 2016 Mar 2. No abstract available. PMID 26947385
- [Background] Schnittger I, Boyd JH, Tremmel JA. A Step Back in the Diagnosis and Management of Myocardial Bridging. Ann Thorac Surg. 2020 Jun;109(6):1950. doi: 10.1016/j.athoracsur.2019.09.051. Epub 2019 Nov 7. No abstract available. PMID 31706871
- [Background] Parikh RV, Pargaonkar V, Ball RL, Kobayashi Y, Kimura T, Yeung AC, Cooke JP, Tremmel JA. Asymmetric dimethylarginine predicts impaired epicardial coronary vasomotion in patients with angina in the absence of obstructive coronary artery disease. Int J Cardiol. 2020 Jan 15;299:7-11. doi: 10.1016/j.ijcard.2019.07.062. Epub 2019 Jul 19. PMID 31416658
- [Background] Nishikii-Tachibana M, Pargaonkar VS, Schnittger I, Haddad F, Rogers IS, Tremmel JA, Wang PJ. Myocardial bridging is associated with exercise-induced ventricular arrhythmia and increases in QT dispersion. Ann Noninvasive Electrocardiol. 2018 Mar;23(2):e12492. doi: 10.1111/anec.12492. Epub 2017 Sep 18. PMID 28921787
- [Background] Boyd JH, Pargaonkar VS, Scoville DH, Rogers IS, Kimura T, Tanaka S, Yamada R, Fischbein MP, Tremmel JA, Mitchell RS, Schnittger I. Surgical Unroofing of Hemodynamically Significant Left Anterior Descending Myocardial Bridges. Ann Thorac Surg. 2017 May;103(5):1443-1450. doi: 10.1016/j.athoracsur.2016.08.035. Epub 2016 Oct 13. PMID 27745841
- [Background] Forsdahl SH, Rogers IS, Schnittger I, Tanaka S, Kimura T, Pargaonkar VS, Chan FP, Fleischmann D, Tremmel JA, Becker HC. Myocardial Bridges on Coronary Computed Tomography Angiography - Correlation With Intravascular Ultrasound and Fractional Flow Reserve. Circ J. 2017 Nov 24;81(12):1894-1900. doi: 10.1253/circj.CJ-17-0284. Epub 2017 Jul 7. PMID 28690285
- [Background] Yamada R, Tremmel JA, Tanaka S, Lin S, Kobayashi Y, Hollak MB, Yock PG, Fitzgerald PJ, Schnittger I, Honda Y. Functional Versus Anatomic Assessment of Myocardial Bridging by Intravascular Ultrasound: Impact of Arterial Compression on Proximal Atherosclerotic Plaque. J Am Heart Assoc. 2016 Apr 20;5(4):e001735. doi: 10.1161/JAHA.114.001735. PMID 27098967
- [Background] Pargaonkar VS, Tremmel JA, Schnittger I, Khandelwal A. Effect of ranolazine on symptom and quality of life in patients with angina in the absence of obstructive coronary artery disease: A case control study. Int J Cardiol. 2020 Jun 15;309:8-13. doi: 10.1016/j.ijcard.2020.02.014. Epub 2020 Feb 6. PMID 32220488
- [Background] Kobayashi Y, Fearon WF, Honda Y, Tanaka S, Pargaonkar V, Fitzgerald PJ, Lee DP, Stefanick M, Yeung AC, Tremmel JA. Effect of Sex Differences on Invasive Measures of Coronary Microvascular Dysfunction in Patients With Angina in the Absence of Obstructive Coronary Artery Disease. JACC Cardiovasc Interv. 2015 Sep;8(11):1433-1441. doi: 10.1016/j.jcin.2015.03.045. PMID 26404195
- [Background] Pargaonkar VS, Lee JH, Chow EKH, Nishi T, Ball RL, Kobayashi Y, Kimura T, Lee DP, Stefanick ML, Fearon WF, Yeung AC, Tremmel JA. Dose-Response Relationship Between Intracoronary Acetylcholine and Minimal Lumen Diameter in Coronary Endothelial Function Testing of Women and Men With Angina and No Obstructive Coronary Artery Disease. Circ Cardiovasc Interv. 2020 Apr;13(4):e008587. doi: 10.1161/CIRCINTERVENTIONS.119.008587. Epub 2020 Apr 13. PMID 32279562
- See also: Women's Heart Health at Stanford homepage — https://stanfordhealthcare.org/medical-clinics/womens-heart-health.html